CLINICAL TRIAL: NCT03736031
Title: With Love: Using Promotoras for a Hispanic Community Palliative Care Intervention - A Pilot Study (Promotora Palliative)
Brief Title: With Love: Using Promotoras for a Hispanic Community Palliative Care Promotora Palliative Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University Health Sciences Center, El Paso (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: E18031
Record Dates: First submitted 2018-04-04; First posted 2018-11-08 (Actual); Results first posted 2020-10-26 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-10

CONDITIONS: Palliative Care
Keywords: cancer
MeSH Terms: conditions — Neoplasms | interventions — Methods

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Promotora) (Experimental): The intervention group will have three face-to-face meetings with the promotora. Participant will continue to receive the standard of care for his or her oncologic diagnosis as determined by his or her treating oncologist over the course of the study. During the study period, all participants will complete baseline, interim and exit surveys covering demographics, quality of life and pain management. Information pertaining to hospitalizations and emergency room visits will be obtained from their medical records and public health records.
  Interventions: Behavioral: Intervention (Promotora)
- Self-Education (Control) (No Intervention): Participant will receive the standard of care for his or her oncologic diagnosis as determined by his or her treating oncologist over the course of the study. During the study period, all participants will complete baseline, interim and exit surveys covering demographics, quality of life and pain management. Information pertaining to hospitalizations and emergency room visits will be obtained from their medical records and public health records.

INTERVENTIONS:
Behavioral: Intervention (Promotora) — If the patient is in the intervention group, the promotora will call the patient in order to invite them to a meeting. Meetings will be arranged by the promotora and the patients. A total of 2 group meetings will be required by all participants and 1 family meeting.
  Arms: Intervention (Promotora)

SUMMARY:
Despite being strongly recommended, the integration of palliative care in oncology has not been widely adopted. Very few people have access to comprehensive palliative care. Access is even lower in rural and Hispanic communities. Even in communities with access, uptake is often low due to a lack of education on the part of both patients and providers regarding palliative care. This study aims to use an innovative approach to provide quality palliative care to oncology Hispanic patients by using community health workers also known as promotoras.

DETAILED DESCRIPTION:
Palliative care has been highly recommended to be an integral part of oncology yet very few people have access to comprehensive palliative care. Access is even lower in rural, low socio-economic and Hispanic communities. Palliative care has been shown to decrease healthcare costs. This study will use an innovative approach to provide quality palliative care to gynecology-oncology Hispanic patients by using community health workers also known as promotoras. The promotora model has been shown to be successful in several behavioral modification programs. The investigators aim to use promotoras to deliver a comprehensive and culturally sensitive educational intervention that covers self-care in the presence of cancer, advance directives, pain management, and care taker awareness. The goal of the intervention will be to decrease number of emergency department visits and hospital admissions of patients with advanced cancer, and increase the rate of completion of advanced directives, as well as improve overall quality of life (as measured by standardized scales) when comparing the intervention group vs. the control (usual care) group. The investigators will additionally assess the cost effectiveness of this intervention.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 years or older
* Must be a Texas Tech University Health Sciences Center El Paso (TTUHSC El Paso) or University Medical Center (UMC) El Paso patient
* Must be Hispanic
* Must have a cancer diagnosis

Exclusion Criteria:

* Under 17 years of age
* Not Hispanic
* Is not a patient of UMC or TTUHSC El Paso

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2018-05-08 (Actual); Primary Completion 2019-10-04 (Actual); Study Completion 2020-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christina Bracamontes, MS, Study Director — Texas Tech University HSC El Paso
Locations (1):
- Texas Tech University Health Sciences Center El Paso, El Paso, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at an academic medical center between May 8, 2018 and August 15, 2019.
Pre-assignment Details: Participant enrollment and randomization occured at the same time. There were no enrolled participants excluded from the study before assignment to groups.
Period: Overall Study
Arm/Group | Intervention (Promotora) | Self-Education (Control)
Started | 56 | 46
Completed | 24 | 40
Not Completed | 32 | 6
Not completed — Death | 2 | 4
Not completed — Lost to Follow-up | 21 | 2
Not completed — Withdrawal by Subject | 9 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention (Promotora) | Self-Education (Control) | Total
Number analyzed (Participants) | 56 | 46 | 102
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.28 (11.79) | 50.7 (11.4) | 52.09 (11.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 10 | 58
  Male | 8 | 36 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 56 | 46 | 102
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 56 | 46 | 102
Education [Count of Participants; unit: Participants]
  No Schooling | 2 | 1 | 3
  Primary School | 10 | 7 | 17
  High School | 24 | 26 | 50
  College | 10 | 3 | 13
  Vocational School | 4 | 3 | 7
  University, College | 6 | 6 | 12
Marital Status [Count of Participants; unit: Participants]
  Married | 25 | 29 | 54
  Single, never married | 11 | 7 | 18
  Divorced/ separated | 20 | 8 | 28
  Widowed | 0 | 2 | 2
Pain [Count of Participants; unit: Participants] — Population: All questions were voluntary. If a participant refused to answer, they were able to skip the question.
  Participants
    Head: number analyzed (Participants) | 50 | 45 | 95
    Head | 2 | 9 | 11
    Chest: number analyzed (Participants) | 49 | 45 | 94
    Chest | 2 | 4 | 6
    Abdomen: number analyzed (Participants) | 50 | 45 | 95
    Abdomen | 11 | 11 | 22
    Wrist: number analyzed (Participants) | 50 | 46 | 96
    Wrist | 4 | 7 | 11
    Knees: number analyzed (Participants) | 50 | 45 | 95
    Knees | 10 | 12 | 22
    Neck: number analyzed (Participants) | 50 | 45 | 95
    Neck | 5 | 4 | 9
    Upper Back: number analyzed (Participants) | 50 | 45 | 95
    Upper Back | 7 | 4 | 11
    Lower Back: number analyzed (Participants) | 50 | 45 | 95
    Lower Back | 9 | 6 | 15
    Upper Arms/ Shoulders: number analyzed (Participants) | 51 | 45 | 96
    Upper Arms/ Shoulders | 6 | 7 | 13

OUTCOME MEASURES:

1. Primary Outcome: Patient Health Questionnaire - 9 (PHQ-9)
Description: Patient Health Questionnaire -9 (PHQ-9); the score can range from 0 - 27; the lower score indicates a better outcome
Time Frame: The PHQ-9 was administered at baseline and then again about six weeks later when study participation is completed..
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention (Promotora) | Self-Education (Control)
Number analyzed (Participants) | 26 | 41
score on a scale
  Baseline | 5.23 (4.7) | 8.83 (6.72)
  Study Completion | 6.77 (6.84) | 7 (5.89)
Statistical Analysis 1: Comparison: Intervention (Promotora) vs Self-Education (Control); Test type: Superiority; p = 0.09, two-sample independent t-test; An alpha of 0.05 was used

2. Primary Outcome: Functional Assessment of Chronic Illness Therapy - Palliative Care (FACIT-Pal)
Description: Functional Assessment Chronic Illness Therapy (FACIT)-Palliative care (Pal), score range 0-184, a higher score means a better outcome.
Time Frame: The FACIT-Pal was administered at baseline and then again about six weeks later when study participation is completed.
Population: Data was only analyzed for participants who completed both the survey at both timepoints (baseline and completion).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention (Promotora) | Self-Education (Control)
Number analyzed (Participants) | 26 | 41
score on a scale
  Baseline | 138.93 (22.95) | 126.43 (27.38)
  Study Completion | 134.04 (45.65) | 119.17 (40.39)
Statistical Analysis 1: Comparison: Intervention (Promotora) vs Self-Education (Control); Test type: Superiority; p = 0.81, two-sample independent t-test; An alpha of 0.05 was used

3. Secondary Outcome: Emergency Department Visits
Description: Frequency of visits will be analyzed as an intent-to-treat analysis
Time Frame: six weeks after enrollment
Measure: Mean (Standard Deviation); unit: visits
Arm/Group | Intervention (Promotora) | Self-Education (Control)
Number analyzed (Participants) | 56 | 46
visits | 1.05 (1.73) | 1.39 (1.74)
Statistical Analysis 1: Comparison: Intervention (Promotora) vs Self-Education (Control); Test type: Superiority; p = 0.33, t-test, 2 sided

4. Secondary Outcome: Intensive Care Unit Admissions
Description: Frequency of visits will be analyzed as an intent-to-treat analysis
Time Frame: six weeks after enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention (Promotora) | Self-Education (Control)
Number analyzed (Participants) | 56 | 46
Participants | 2 | 1
Statistical Analysis 1: Comparison: Intervention (Promotora) vs Self-Education (Control); Test type: Superiority; p = 1.0, Fisher Exact

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Intervention (Promotora) | Self-Education (Control)
All-Cause Mortality (participants affected / at risk) | 2/56 | 4/46
Serious Adverse Events (participants affected / at risk) | 2/56 | 1/46
Other Adverse Events (participants affected / at risk) | 27/56 | 21/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention (Promotora) (N=56) | Self-Education (Control) (N=46)
Hospital admission (General disorders) | 2 | 1 — This event was not related to the intervention.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention (Promotora) (N=56) | Self-Education (Control) (N=46)
Nausea (Gastrointestinal disorders) | 14 | 9 — This event was not related to the intervention.
Pain (General disorders) | 10 | 9 — This event was not related to the intervention.
Swelling (Blood and lymphatic system disorders) | 3 | 3 — This event was not related to the intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2019-03-28): https://cdn.clinicaltrials.gov/large-docs/31/NCT03736031/Prot_002.pdf
  • Informed Consent Form (2018-10-16): https://cdn.clinicaltrials.gov/large-docs/31/NCT03736031/ICF_003.pdf
  • Statistical Analysis Plan (2019-03-28): https://cdn.clinicaltrials.gov/large-docs/31/NCT03736031/SAP_004.pdf